CLINICAL TRIAL: NCT06948799
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Immunogenicity of STSP-0902 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Tolerability of Multiple Dose of STSP-0902 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSP-0902-01-002
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Oligozoospermia
MeSH Terms: conditions — Oligospermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low dose of STSP-0902 subcutaneous injection or dose-matched placebo (First cohort) (Experimental): 12 subjects will be randomized to receive lowest dose of STSP-0902 subcutaneous injection or dose-matched placebo (First cohort)
  Interventions: Drug: STSP-0902 injection; Drug: Placebo
- middle dose of STSP-0902 subcutaneous injection or dose-matched placebo (Second cohort) (Experimental): 12 subjects will be randomized to receive middle dose of STSP-0902 subcutaneous injection or dose-matched placebo (Second cohort)
  Interventions: Drug: STSP-0902 injection; Drug: Placebo
- high dose of STSP-0902 subcutaneous injection or dose-matched placebo (Third cohort) (Experimental): 12 subjects will be randomized to receive high dose of STSP-0902 subcutaneous injection or dose-matched placebo (Third cohort)
  Interventions: Drug: STSP-0902 injection; Drug: Placebo
- higher dose of STSP-0902 subcutaneous injection or dose-matched placebo (fourth cohort) (Experimental): 12 subjects will be randomized to receive high dose of STSP-0902 subcutaneous injection or dose-matched placebo (fourth cohort)
  Interventions: Drug: STSP-0902 injection; Drug: Placebo

INTERVENTIONS:
Drug: STSP-0902 injection — Subjects will receive the administration dose on Day 1 following protocol requirements
Drug: Placebo — Subjects will receive the administration dose on Day 1 following protocol requirements

SUMMARY:
This is a Phase 1b, randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of STSP-0902

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers, aged between 18 and 50 years inclusive, with a body weight of at least 50.0 kg, and a body mass index (BMI) between 19.0 and 28.0 kg/m² inclusive, and whose two routine semen analysis results during the screening period meet the criteria of sperm concentration of less than 15 million and/or percentage of progressively motility sperm of less than 32%.
2. Participants (including the partners of the participants) must use effective non-drug contraceptive measures during the trial period and for four months after the end of administration, and must not have plans for pregnancy or sperm donation.
3. Participants should avoid high temperature environments during the trial, including saunas, steam baths, hot baths, hot springs, and the use of electric blankets.
4. Participants must give informed consent to this study before the study and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Participants with a history of severe diseases, including but not limited to conditions affecting the skeletal, neuropsychiatric, cardiovascular, hematologic, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immune, and reproductive systems (such as reproductive system infectious diseases, varicocele, reproductive tract obstruction, etc., except for oligoasthenzoospermia), as judged by the investigator, may endanger the safety of the participant or affect the study results.
2. Participants who have planned to receive treatments related to oligoasthenzoospermia, such as zinc sulfate, levocarnitine, escin, or pancreatic kallikrein, within 3 months prior to screening or during the trial period.
3. Participants with a history of treatment with nerve growth factor-like drug therapy (such as mouse nerve growth factor for injection) within 3 months prior to screening.
4. Participants who have undergone any major surgery within 3 months prior to screening or have surgery planned during the trial period.
5. Participants who have experienced a fever exceeding 38 ℃ within 1 month prior to screening
6. Pre-enrollment physical examination, electrocardiogram, vital signs, laboratory tests, and results of all tests related to the trial (except oligoasthenzoospermia), with abnormalities judged clinically significant by the investigator.
7. Participants who are allergic to any component of the experimental drug or biological agent, or who, in the judgment of the investigator, are at risk of allergy as a result of participation in the study.
8. Participants who are positive for any one of the hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, and HIV antigen/antibody combination test (primary screening).
9. Tattoos at the injection site or other skin conditions that interfere with observation of the skin.
10. Participants who have smoked more than 5 cigarettes per day or an equivalent amount of tobacco in the 3 months prior to screening.
11. Participants with frequent alcohol consumption within 6 months prior to screening, i.e., more than 2 units of alcohol per day (1 unit = 360 ml of beer or 45 ml of spirits of 40% alcohol by volume or 150 ml of wine); or those with a positive alcohol breath test.
12. Participants who have habitual consumption of more than 5 cups of coffee, tea or cola, etc. per day (150 ml and above per cup) in the 3 months prior to screening.
13. Participants who have a history of drug abuse within 1 year prior to screening or have a positive urine drug test.
14. Participants who have participated in blood donation within 3 months prior to screening with a total blood donation of ≥ 400 mL or total blood loss of ≥ 400 mL, or who have history of blood transfusion within 4 weeks prior to enrollment.
15. Participants who have taken any investigational product or participated in any clinical trial of drug, devices or vaccines intervention within 3 months prior to screening.
16. Vaccination within 1 month prior to screening or scheduled to be administered during the study period up to 2 months after completion of the study.
17. Participants who have used any prescription, over-the-counter medications or herbal remedies within 14 days prior to screening.
18. Participants with a history of fear of needles and homophobia.
19. Participants with other factors that are not suitable for participation in this study as judged by the investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-related adverse events as assessed by CTCAE 5.0. | 85 days
  To evaluate the safety and tolerability of STSP-0902 injection in healthy adult subjects

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) | From pre-dose up to 21 days post last dose
  To evaluate the pharmacokinetics (PK) of STSP-0902
Area under the plasma concentration-time curve (AUC0-t) | From pre-dose up to 21 days post last dose
  To evaluate the pharmacokinetics (PK) of STSP-0902
Area under the curve from time 0 extrapolated to infinite time (AUC0-∞) | From pre-dose up to 21 days post last dose
  To evaluate the pharmacokinetics (PK) of STSP-0902
Time to peak Concentration (Tmax) | From pre-dose up to 21 days post last dose
  To evaluate the pharmacokinetics (PK) of STSP-0902
Elimination Phase Half-life (t1/2) | From pre-dose up to 21 days post last dose
  To evaluate the pharmacokinetics (PK) of STSP-0902
apparent oral clearance (CL/F) | From pre-dose up to 21 days post last dose
  To evaluate the pharmacokinetics (PK) of STSP-0902
Anti-drug antibody(ADA) | From pre-dose up to 56 days post last dose
  To evaluate the immunogenicity of STSP-0902

OTHER OUTCOMES:
Tests for sex hormones (including follicle-stimulating hormone, luteinizing hormone, estradiol, progesterone, testosterone and prolactin), norepinephrine and methoxy norepinephrine | 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Kai Hong, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China